CLINICAL TRIAL: NCT02915679
Title: Pain Perception in Suicidal Behavior Vulnerability
Acronym: DOCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 9185; 2013-A01029-36 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-08-01; First posted 2016-09-27 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Episode
Keywords: Suicidal behavior; psychological and social pain; physical pain; pain perception
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study participant (Other): All the participants performed blood sample for genetic purpose, psychiatric assessment and pain investigation:
  * 81 depressed patients admitted after a recent suicidal act (<8 days)
  * 81 depressed subjects with a past history of suicidal act (>1month)
  * 80 depressed subjects without any personal history of suicidal behaviour
  Interventions: Other: Blood sample for genetic purpose, psychiatric assessment and pain investigation

INTERVENTIONS:
Other: Blood sample for genetic purpose, psychiatric assessment and pain investigation — All the participant will performed the same evaluation and blood analysis:
  * A clinical assessment by psychiatrics assessing psychiatric disorder and suicidal behavior
  * Thermal stimulation for pain assessment
  * Computer game named Cyberball: test of social exclusion
  * Self report questionnaire for the assessment of reject sensitivity, relationship style, impulsivity, childhood trauma.
  * Routine blood sampling

SUMMARY:
In France, almost 1 death on 50 is a suicide. The suicide occurs in unbearable psychic pain where mental trouble has a major influence. It is classified as preventable mortality. According to interpersonal psychological theory of suicide, the repeated exposition to stressful and painful events (as physical abuse) would facilitate suicide attempt through the increased pain tolerance. The social pain (or psychical pain on the broader sense) and physical pain are closely linked.

The investigators hypothesize that the measure of painful perception will be significantly superior on suicidals attempters compared to non-attempters. It will be the case for recent suicide attempters and former suicide attempters, suggesting a suicidal vulnerability trait. Moreover, the investigators expect that social distress induced by a social exclusion paradigm will be significantly superior on suicide attempters compared to non-attempters.

The aim of the study is to investigate the physical and psychic pain on depressed subjects with or without history of suicide attempts.

After a clinical evaluation (psychiatric symptomatology, personality trait, suicidal dimension), subjects will be submitted to a painful thermic stimulation and will participate at a computer test of social exclusion (named Cyberball).

DETAILED DESCRIPTION:
242 depressed patients ( 81 recent suicide attempters, 81 former suicide attempters, 80 non-attempters)

First visit : clinical assessment Second visit : pain evaluation and blood sample (from one day to a week maximum after the first visit).

ELIGIBILITY:
Inclusion criteria:

* aged by 18 years old
* came from West Europe, excepted Basque and Sardinian (because of genetics analysis)
* main diagnosis of major depressive episode (DSM V criteria)
* not having take antalgics in the 24 hours before assessment
* received a minimal psychotrope treatment (clinician evaluation)
* Able to understand nature, aims, methodology of the study
* Agree to cooperate in clinical and biological assessment
* Having signed informed consent

Specific inclusion criteria :

81 recent suicide attempters (being hospitalised for suicidal attempts and having realised a suicide attempts 8 days before inclusion) 81 former suicide attempters (having realised in his lifetime a suicide attempt, one month before inclusion)

Exclusion criteria:

* Current diagnosis of manic, hypomanic or alcohol dependance or substance abuse in the last 6 months, or diagnosis of schizophrenia or schizoaffective disorder in his lifetime
* Current algic and chronic neurologic disease
* Current or actual treatment by tricyclic antidepressant and Serotonin and norepinephrine reuptake inhibitors(SNRIs)
* Pregnancy
* Patients on protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-06-17; Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Pain tolerance reported by the patient | During thermal stimulation
  temperature measured when the subject will perceive as intolerable the pain following a painful stimulation performed using a thermode

SECONDARY OUTCOMES:
Pain intensity reported by the patient | During thermal stimulation
  comparison between the three groups of the pain intensity (assessed by likert scale) at constant temperature (43 ° C)
Pain threshold reported by the patient | During thermal stimulation
  comparison between the three groups of the pain threshold (temperature perceived as painful)
Temperature assessed at 4/10 on likert scale | During thermal stimulation performed at the inclusion
  comparison between the three groups of the temperature assessed at 4/10 on a visual analogic painful scale, kinetics of pain intensity by visual analog scale (VAS) scale.
Kinetics of pain intensity | During thermal stimulation performed at the inclusion
  comparison between the three groups of kinetics of pain intensity by visual analog scale (VAS) scale.
Social distress perception assessed by social distress questionnaire | At V2 (one week maximum after the inclusion)
  comparison between the three groups of the score of social distress scale after cyberball game
Social distress perception assessed by the Rejection Sensitivity Questionnaire (RSQ) | At the inclusion
  comparison between the three groups of the score of social distress scale after cyberball game
Social rejection sensitivity assessed by the Rejection Sensitivity Questionnaire (RSQ) | At the inclusion
  comparison between the three groups of the score of social rejection sensitivity by RSQ
Psychological pain intensity | At V2 (one week maximum after the inclusion)
  comparison between the three groups of the score of psychological pain intensity assessed by VAS scale.
Measure of cardiac frequency in response to thermal pain | At V2 (one week maximum after the inclusion)
  comparison between the three groups of the cardiac frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier Hospital University, Montpellier, France

IPD SHARING:
Plan to Share IPD: No